Title: Acceptability/Feasibility Testing of SCAR

**Document Date: 4/21/2021** 

## **Data Analytic Plan**

Consistent with recommendations for determining acceptability and feasibility in the context of intervention development, multiple program aspects will be evaluated with the aim of refining SCAR for larger-scale implementation. Feasibility of SCAR will be indexed via participant retention, average homework completion, and percentage of EMA sessions completed. The EMI will be considered feasible if > 80% of the EMA sessions are completed by > 80% of participants, as done in previous studies (LaFreniere & Newman, 2016; Lucas-Thompson et al., 2019). Acceptability of SCAR will be measured using the CSQ-8, an 8-item measure that assesses general program satisfaction. An average CSQ-8 rating of > 3 (on a 4-point scale) will provide support for the acceptability of this intervention. Participant feedback will also be used to further examine potential reasons for drop-out and non-adherence to inform our future study. Therapist fidelity scores for the individual session will be assessed as the percentage of the content delivered. Interrater reliability for fidelity and competence will be assessed using intraclass correlation coefficients.

Secondary analyses will be conducted to determine the effect of the SCAR intervention on social anxiety and anxiety sensitivity social concerns. Means and standard deviations for outcomes will be calculated at each assessment, including change scores and correlations across timepoints. We expect large standard errors due to sample size. Distribution of scores will be examined to better evaluate how to analyze these data in future studies (e.g., categorizing vs. continuous). For continuous outcomes, Hedge's g will be calculated to identify a range of the pre-post effect size. Although such calculations are of limited benefit in determining the effect of the intervention, they can be helpful in identifying outcomes for which the intervention may be less effective. Correlations among baseline variables will be calculated to assess the potential for

variables to be stratified or included as covariates in a larger trial. This may also be useful in identifying potential moderators and mediators for a future larger trial. For data quality and handling of missing data, descriptive statistics will help identify outliers.